CLINICAL TRIAL: NCT06480786
Title: Spinal Cord Stimulation for Patients With Painful Diabetic Neuropathy and Peripheral Arterial Disease: Mechanistic Insights From a Single-center, Randomized, Blinded, Sham-controlled Cross-over Proof-of-concept Trial
Brief Title: SCS for Patient With Painful Diabetic Neuropathy and Peripheral Arterial Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Nevro Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0623-24-FB
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Arterial Disease; Painful Diabetic Neuropathy; Diabetes Mellitus, Type 2; Chronic Pain; Spinal Cord Stimulation; Chronic Pain Syndrome; Limb Pain
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetic Neuropathies; Diabetes Mellitus, Type 2; Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: 1:1 cross over design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Spinal Cord Stimulation (Experimental): Therapeutic spinal cord stimulation titrated at 12 weeks post operative at standard clinical practice.
  Interventions: Device: Spinal cord stimulation
- Sham Stimulation (Sham Comparator): Sub-threshold low frequency spinal cord stimulation to provide no analgesic benefit but serve as a sham control.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Spinal cord stimulation — active spinal cord stimulation
  Arms: Active Spinal Cord Stimulation
Device: Sham stimulation — Sham stimulation
  Arms: Sham Stimulation

SUMMARY:
Peripheral arterial disease (PAD) affects over 230 million adults worldwide and is a highly morbid, costly, and disabling condition. Ischemic leg pain drives disability in PAD patients and results from oxygen supply-demand mismatch, autonomic dysfunction, and muscle breakdown. This leg pain, which is unresponsive to traditional pharmacotherapy, limits the patient's tolerance to exercise, which is an important disease-modifying intervention. Spinal cord stimulation is a well-established therapy for medically intractable pain, including painful diabetic neuropathy (PDN) and ischemic pain, but is not part of the standard-of-care for PAD despite limited promising clinical data. Early studies used first-generation, tonic stimulation devices, but with these it was impossible to perform sham-controlled trials to test the treatment. Since then, new types of waveform treatments, including high-frequency spinal cord stimulation (SCS), have been shown to be more effective in the treatment of intractable pain. While high-frequency SCS is approved for PDN treatment, it has never been tested in the treatment of claudication pain from PAD.

This study will enroll up to 15 participants between the ages of 19 and 89 who have PAD and PDN and are successfully implanted with a permanent SCS. Twelve weeks after SCS implantation, participants will receive two weeks of stimulation and two weeks of sham intervention, in random starting order. Blood flow, blood pressure, skin oxygen levels, and participant reported pain int the lower extremities will be assessed before SCS implantation, 12 weeks after SCS implantation and during each of the treatment periods. Participants will also complete a quality of life survey at the same time points. Comparisons of these measurements with the baseline and post-implantation measurements to determine the effects of SCS.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) affects over 230 million adults worldwide and is a highly morbid, costly, and disabling condition. Ischemic leg pain drives disability in PAD patients and results from oxygen supply-demand mismatch, autonomic dysfunction, and muscle breakdown. This leg pain, which is unresponsive to traditional pharmacotherapy, limits the patient's tolerance to exercise, which is an important disease-modifying intervention. Spinal cord stimulation is a well-established therapy for medically intractable pain, including painful diabetic neuropathy (PDN) and ischemic pain, but is not part of the standard-of-care for PAD despite limited promising clinical data. Early studies used first-generation, tonic stimulation devices, but with these it was impossible to perform sham-controlled trials to test the treatment. Since then, new types of waveform treatments, including high-frequency spinal cord stimulation (SCS), have been shown to be more effective in the treatment of intractable pain. While high-frequency SCS is approved for PDN treatment, it has never been tested in the treatment of claudication pain from PAD.

This study will enroll up to 15 participants between the ages of 19 and 89 who have PAD (ankle-brachial index under 0.90 or vascular imaging, and experience pain from walking with a pain level of at least 6 cm for at least 3 months )and PDN and who meet inclusion criteria for permanent spinal cord stimulator (SCS) placement. Participants must also have diabetes with symptoms of neuropathy, have a starting pain level of at least 5 cm on a visual pain scale and Vascular Quality of Life Questionnaire score of 5.5 or less.

The study begins with an initial evaluation visit, then a follow-up visit 12 weeks after permanent SCS implantation and optimization. Participants will then be randomized to start in the SCS group or the sham intervention group. Each of these interventions will be conducted for two weeks, then participants will switch to the other intervention in a cross over design. Blood flow, blood pressure, skin oxygen levels, and participant reported pain int the lower extremities will be assessed before SCS implantation, 12 weeks after SCS implantation and during each of the treatment periods. Participants will also complete a quality of life survey at the same time points. Comparisons of these measurements with the baseline and post-implantation measurements to determine the effects of SCS. The study intervention lasts for 4 weeks, after which participants will return to standard SCS care.

ELIGIBILITY:
Inclusion Criteria:

* 19 years to 89 years old
* Diagnosed diabetes mellitus
* Signs or symptoms of neuropathy and maximum baseline visual-analog pain scale ≥ 5 cm and peripheral arterial disease (diagnosed by ankle-brachial index < 0.90 or vascular imaging studies) with claudication and exertion-induced visual-analog pain scale ≥ 6 cm for a minimum of 3 months
* Successful spinal cord stimulator (SCS) trial (>50% relief of chronic lower extremity pain) and will have a new permanent SCS placed prior to study intervention

Exclusion Criteria:

* Uncontrolled psychological or psychiatric disorder
* Inability to hold antithrombotic therapy per the American Society of Regional Anesthesia guidelines
* Non-healing wounds
* Gangrene
* Critical limb ischemia
* Prior lower extremity amputation
* Inability to adhere to study follow-up
* Mechanical spine instability based on flexion/extension radiographs of the lumbar spine
* Prior or current spinal cord stimulator implant

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
High-frequency Spinal Cord Stimulation Effect on Analgesia | Baseline, 12 week follow-up after permanent spinal cord simulator, week 14 intervention #1 , week 16 intervention #2
  The visual analogue scale (VAS) will be used by participants to report lower extremity pain during interventions. The VAS score is a10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
High-frequency Spinal Cord Stimulation Effect on Quality of Life | Baseline, 12 week follow up after permanent spinal cord simulator, week 14 intervention #1 , week 16 intervention #2
  Quality of life changes from high-frequency high-frequency spinal cord stimulation (SCS) will be measured by the Vascular Quality of Life Questionnaire (VASCUQOL). This instrument has 25 questions covering pain, symptoms, activities, social, and emotional. Each question has seven responses from 1 (worst) to 7 (best).
High-frequency Spinal Cord Stimulation Effect on Blood Flow | Baseline, 12 week follow up after permanent spinal cord simulator, week 14 intervention #1 , week 16 intervention #2
  Changes in blood flow from high-frequency spinal cord stimulation (SCS) will measure lower extremity capillary digit blood flow flow by laser speckle imaging.
High-frequency Spinal Cord Stimulation Effect on Autonomic Control | Baseline, 12 week follow-up after permanent spinal cord simulator, week 14 intervention #1 , week 16 intervention #2
  Changes in autonomic control from high-frequency spinal cord stimulation (SCS) will measure sympathetic vasomotion by volume-clamp method on digits of the hand and laser speckle imaging on the lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pellegrino, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersen EA, Stauss TG, Scowcroft JA, Brooks ES, White JL, Sills SM, Amirdelfan K, Guirguis MN, Xu J, Yu C, Nairizi A, Patterson DG, Tsoulfas KC, Creamer MJ, Galan V, Bundschu RH, Paul CA, Mehta ND, Choi H, Sayed D, Lad SP, DiBenedetto DJ, Sethi KA, Goree JH, Bennett MT, Harrison NJ, Israel AF, Chang P, Wu PW, Gekht G, Argoff CE, Nasr CE, Taylor RS, Subbaroyan J, Gliner BE, Caraway DL, Mekhail NA. Effect of High-frequency (10-kHz) Spinal Cord Stimulation in Patients With Painful Diabetic Neuropathy: A Randomized Clinical Trial. JAMA Neurol. 2021 Jun 1;78(6):687-698. doi: 10.1001/jamaneurol.2021.0538. PMID 33818600
- [Background] Pellegrino PR, Zucker IH, Chatzizisis YS, Wang HJ, Schiller AM. Quantification of Renal Sympathetic Vasomotion as a Novel End Point for Renal Denervation. Hypertension. 2020 Oct;76(4):1247-1255. doi: 10.1161/HYPERTENSIONAHA.120.15325. Epub 2020 Aug 24. PMID 32829663
- [Background] Al-Kaisy A, Palmisani S, Pang D, Sanderson K, Wesley S, Tan Y, McCammon S, Trescott A. Prospective, Randomized, Sham-Control, Double Blind, Crossover Trial of Subthreshold Spinal Cord Stimulation at Various Kilohertz Frequencies in Subjects Suffering From Failed Back Surgery Syndrome (SCS Frequency Study). Neuromodulation. 2018 Jul;21(5):457-465. doi: 10.1111/ner.12771. Epub 2018 Apr 2. PMID 29608229
- [Background] Kretzschmar M, Okaro U, Schwarz M, Reining M, Lesser T. Spinal Neuromodulation for Peripheral Arterial Disease of Lower Extremities: A Ten-Year Retrospective Analysis. Neuromodulation. 2024 Oct;27(7):1240-1250. doi: 10.1016/j.neurom.2023.10.186. Epub 2024 Jan 1. PMID 38165292
- [Background] Piedade GS, Vesper J, Reichstein D, Dauphin AK, Damirchi S. Spinal cord stimulation in non-reconstructable critical limb ischemia: a retrospective study of 71 cases. Acta Neurochir (Wien). 2023 Apr;165(4):967-973. doi: 10.1007/s00701-022-05448-8. Epub 2023 Jan 4. PMID 36598544
- [Background] Klinkova A, Kamenskaya O, Ashurkov A, Murtazin V, Orlov K, Lomivorotov VV, Karaskov A. The Clinical Outcomes in Patients with Critical Limb Ischemia One Year after Spinal Cord Stimulation. Ann Vasc Surg. 2020 Jan;62:356-364. doi: 10.1016/j.avsg.2018.12.093. Epub 2019 Feb 22. PMID 30802587
- [Background] Deogaonkar M, Zibly Z, Slavin KV. Spinal cord stimulation for the treatment of vascular pathology. Neurosurg Clin N Am. 2014 Jan;25(1):25-31. doi: 10.1016/j.nec.2013.08.013. Epub 2013 Oct 5. PMID 24262897
- [Background] Petrakis E, Sciacca V. Prospective study of transcutaneous oxygen tension (TcPO2) measurement in the testing period of spinal cord stimulation in diabetic patients with critical lower limb ischaemia. Int Angiol. 2000 Mar;19(1):18-25. PMID 10853681
- [Background] Chapman KB, Kloosterman J, Schor JA, Girardi GE, van Helmond N, Yousef TA. Objective Improvements in Peripheral Arterial Disease from Dorsal Root Ganglion Stimulation: A Case Series. Ann Vasc Surg. 2021 Jul;74:519.e7-519.e16. doi: 10.1016/j.avsg.2021.01.069. Epub 2021 Feb 4. PMID 33549777
- [Background] De Caridi G, Massara M, David A, Giardina M, La Spada M, Stilo F, Spinelli F, Grande R, Butrico L, de Franciscis S, Serra R. Spinal cord stimulation to achieve wound healing in a primary lower limb critical ischaemia referral centre. Int Wound J. 2016 Apr;13(2):220-5. doi: 10.1111/iwj.12272. Epub 2014 Apr 8. PMID 24712687
- [Background] Cucuruz B, Kopp R, Hampe-Hecht H, Andercou O, Schierling W, Pfister K, Koller M, Noppeney T. Treatment of end-stage peripheral artery disease by neuromodulation. Clin Hemorheol Microcirc. 2022;81(4):315-324. doi: 10.3233/CH-221436. PMID 35466931
- [Background] Cyrek AE, Henn N, Meinhardt F, Lainka M, Pacha A, Paul A, Koch D. Improving Limb Salvage for Chronic Limb-Threatening Ischemia With Spinal Cord Stimulation: A Retrospective Analysis. Vasc Endovascular Surg. 2021 May;55(4):367-373. doi: 10.1177/1538574420985765. Epub 2021 Feb 8. PMID 33550918
- [Background] Petrakis IE, Sciacca V. Does autonomic neuropathy influence spinal cord stimulation therapy success in diabetic patients with critical lower limb ischemia? Surg Neurol. 2000 Feb;53(2):182-8; discussion 188-9. doi: 10.1016/s0090-3019(99)00182-2. PMID 10713199
- [Background] Kilchukov M, Kiselev R, Gorbatykh A, Klinkova A, Murtazin V, Kamenskaya O, Orlov K. High-Frequency versus Low-Frequency Spinal Cord Stimulation in Treatment of Chronic Limb-Threatening Ischemia: Short-Term Results of a Randomized Trial. Stereotact Funct Neurosurg. 2023;101(1):1-11. doi: 10.1159/000527309. Epub 2023 Jan 6. PMID 36617410
- [Background] Abu Dabrh AM, Steffen MW, Asi N, Undavalli C, Wang Z, Elamin MB, Conte MS, Murad MH. Nonrevascularization-based treatments in patients with severe or critical limb ischemia. J Vasc Surg. 2015 Nov;62(5):1330-9.e13. doi: 10.1016/j.jvs.2015.07.069. Epub 2015 Sep 26. PMID 26409842
- [Background] Petrakis IE, Sciacca V. Epidural spinal cord electrical stimulation in diabetic critical lower limb ischemia. J Diabetes Complications. 1999 Sep-Dec;13(5-6):293-9. doi: 10.1016/s1056-8727(99)00061-6. PMID 10765005
- [Background] Mingoli A, Sciacca V, Tamorri M, Fiume D, Sapienza P. Clinical results of epidural spinal cord electrical stimulation in patients affected with limb-threatening chronic arterial obstructive disease. Angiology. 1993 Jan;44(1):21-5. doi: 10.1177/000331979304400104. PMID 8424581
- [Background] Vincenzo S, Kyventidis T. Epidural spinal cord stimulation in lower limb ischemia. Acta Neurochir Suppl. 2007;97(Pt 1):253-8. doi: 10.1007/978-3-211-33079-1_34. PMID 17691384
- [Background] Myklebust JB, Cusick JF, Boerboom LE, Prieto TE, Khan TA. Vascular effects of spinal cord stimulation in the monkey. Stereotact Funct Neurosurg. 1995;64(1):32-9. doi: 10.1159/000098731. PMID 8751312
- [Background] Tedesco A, D'Addato M. Spinal cord stimulation for patients with critical limb ischemia: immediate and long-term clinical outcome from the prospective italian register. Neuromodulation. 2004 Apr;7(2):97-102. doi: 10.1111/j.1094-7159.2004.04013.x. PMID 22151190
- [Background] Horsch S, Claeys L. Epidural spinal cord stimulation in the treatment of severe peripheral arterial occlusive disease. Ann Vasc Surg. 1994 Sep;8(5):468-74. doi: 10.1007/BF02133067. PMID 7811584
- [Background] Broseta J, Barbera J, de Vera JA, Barcia-Salorio JL, Garcia-March G, Gonzalez-Darder J, Rovaina F, Joanes V. Spinal cord stimulation in peripheral arterial disease. A cooperative study. J Neurosurg. 1986 Jan;64(1):71-80. doi: 10.3171/jns.1986.64.1.0071. PMID 3484519